CLINICAL TRIAL: NCT00322491
Title: Treatment With AMD3100 in Non-Hodgkin's Lymphoma and Multiple Myeloma Patients to Increase the Number of Peripheral Blood Stem Cells When Given a Mobilizing Regimen of G-CSF
Brief Title: Mobilization of Stem Cells With AMD3100 (Plerixafor) and G-CSF in Non-Hodgkin's Lymphoma and Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: AnorMED (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-2105
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Results first posted 2010-11-24 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma, Non-Hodgkin; Multiple Myeloma
Keywords: Non-Hodgkin's Lymphoma; Multiple Myeloma; Stem cell mobilization
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Hodgkin's Lymphoma (NHL) (Experimental): Participants with NHL were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Interventions: Drug: G-CSF Plus Plerixafor
- Multiple Myeloma (MM) (Experimental): Participants with MM were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Interventions: Drug: G-CSF Plus Plerixafor

INTERVENTIONS:
Drug: G-CSF Plus Plerixafor — Participants underwent mobilization with G-CSF 10 µg/kg/day for 4 days, administered by subcutaneous injection (SC) injection each morning. On the evening of Day 4, participants received a dose of plerixafor 240 µg/kg, administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF 10 µg/kg and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor (within 60 minutes after administration of G-CSF). Participants continued to receive an evening dose of plerixafor followed the next day by a morning dose of G-CSF and apheresis for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Other Names: AMD3100; Mozobil

SUMMARY:
This study evaluates the safety and efficacy of plerixafor given in addition to granulocyte-colony stimulating factor (G-CSF) for collection of peripheral blood stem cells (PBSCs) for autologous transplantation in patients with non-Hodgkin's lymphoma (NHL) and multiple myeloma (MM). Efficacy outcomes include evaluation of fold increase in circulating CD34+ cells from just before the first plerixafor injection to 10-11 hours post plerixafor (just before apheresis) and assessment of successful polymorphonuclear leukocyte (PMN) engraftment after transplantation. Data from this protocol will assist in the determination of the dosing schedule for future studies.

DETAILED DESCRIPTION:
Participants with NHL and MM who have undergone prior cyto-reductive chemotherapy, are to be autologously transplanted, and meet the inclusion/exclusion criteria are eligible to enter the study. The only change to the standard of care is the addition of plerixafor to a granulocyte colony-stimulating factor (G-CSF) mobilization regimen on the day prior to apheresis. Participants will undergo mobilization with G-CSF (10 mcg/kg each day) and will receive plerixafor (240 mcg/kg) in the evening prior to apheresis. Participants will undergo apheresis for up to 5 consecutive days in order to collect the target number of CD34+ stem cells (≥ 5*10^6 CD34+ cells/kg for either single or tandem transplant). After apheresis, all participants will be treated with high-dose chemotherapy in preparation for transplantation. Participants will be transplanted with cells obtained from the G-CSF and plerixafor mobilization regimen. The increase in CD34+ cells in the peripheral blood from the time of the plerixafor dose to just prior to apheresis and the number of CD34+ cells in the apheresis product will be measured. The number of apheresis sessions required to obtain ≥ 5*10^6 CD34+ cells will also be measured. Success of the transplantation(s) will be evaluated by the time to engraftment of polymorphonuclear leukocytes (PMN) and platelets (PLT). Participants will be followed for durability of their transplant for 12 months following transplantation.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin's lymphoma (NHL) or multiple myoloma (MM) eligible for autologous transplantation
* No more than 3 prior regimens of chemotherapy
* More than 4 weeks since last cycle of chemotherapy. Patient recovered from all acute toxic effects of prior chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell (WBC) count >3.0*10^9/L
* Absolute polymorphonuclear cells (PMN) count >1.5*10^9/L
* Platelet (PLT) count >100*10^9/L
* Serum creatinine <=2.2 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) and total bilirubin <2 x upper limit of normal (ULN)
* Left ventricle ejection fraction >45% by normal echocardiogram or multiple-gated acquisition (MUGA) scan
* Forced expiratory volume of the lung in the first second (FEV1) >60% of predicted or diffusing capacity of the lung for carbon monoxide (DLCO) >45% of predicted
* Negative for human immunodeficiency virus (HIV) type 1
* Women of child bearing potential agreed to use an approved form of contraception.

Exclusion Criteria:

* Patients who have failed previous collections
* Brain metastases or carcinomatous meningitis
* History of ventricular arrhythmias
* A co-morbid condition which, in the view of the investigator, renders the patient at high risk for treatment complications
* A residual acute medical condition resulting from prior chemotherapy
* Acute infection
* Fever (temp >38°C/100.4°F)
* Patients whose actual body weight exceeds 175% of their ideal body weight
* Patients who previously received experimental therapy within 4 weeks of enrolling in this study or who are currently enrolled in another experimental study during the mobilization period
* Positive pregnancy test in female patients
* Lactating females
* Patients of child-bearing potential unwilling to implement adequate birth control.
* Patients who have deterioration of their clinical status or laboratory parameters between the time of enrolment and transplant (such that they no longer meet entry criteria) may be removed from study at the discretion of the treating physician, principal investigator, or sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA School of Medicine, Loa Angeles, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Stiff P, Micallef I, McCarthy P, Magalhaes-Silverman M, Weisdorf D, Territo M, Badel K, Calandra G. Treatment with plerixafor in non-Hodgkin's lymphoma and multiple myeloma patients to increase the number of peripheral blood stem cells when given a mobilizing regimen of G-CSF: implications for the heavily pretreated patient. Biol Blood Marrow Transplant. 2009 Feb;15(2):249-56. doi: 10.1016/j.bbmt.2008.11.028. PMID 19167685

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Started | 23 | 26
Completed | 21 | 24
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.7) | 57.6 (8.1) | 57.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 14 | 16 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23 | 23 | 46
  African-American | 0 | 1 | 1
  Hispanic/Latino | 0 | 1 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Overall Safety Summary of Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with treatment emergent adverse events (TEAEs) collected from Day 1 (start of G-CSF mobilization) to the day before starting chemotherapy (approximately day 38). AEs were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe) and relatedness to study treatment (5 point scale from 'not related' to 'definitely related').
Time Frame: Day 1 to approximately Day 38 (before start of chemotherapy)
Population: Safety population - all participants who received at least 1 dose of plerixafor.
Measure: Number; unit: participants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 23 | 26 | 49
participants
  Participants reporting ≥ 1 Adverse Event | 23 | 26 | 49
  AE Severity (Mild) | 8 | 9 | 17
  AE Severity (Moderate) | 5 | 2 | 7
  AE Severity (Severe) | 10 | 15 | 25
  AE Relationship to Drug (Not Related) | 0 | 4 | 4
  AE Relationship to Drug (Probably Not Related) | 1 | 4 | 5
  AE Relationship to Drug (Possibly Related) | 12 | 5 | 17
  AE Relationship to Drug (Probably Related) | 8 | 11 | 19
  AE Relationship to Drug (Definitely Related) | 2 | 2 | 4

2. Secondary Outcome: Number of Participants Achieving a Two-Fold (Relative) Increase in Peripheral Blood (PB) CD34+ Cells/µL Following the First Dose of Plerixafor
Description: The number of participants mobilized with G-CSF + plerixafor injection who have a ≥ 2-fold increase in CD34+ cells. Fold increase was expressed as a ratio. Fold increase = (pre-apheresis PB CD34+ cells/µL) / (pre-plerixafor dosing PB CD34+ cells/µL)
Time Frame: Days 4-5 (first dose of plerixafor to apheresis)
Population: The intent-to-treat population (defined as participants who received at least 1 dose of plerixafor).
Measure: Number; unit: participants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 23 | 26 | 49
participants
  ≥ 2-fold Increase | 20 | 17 | 37
  < 2-fold Increase | 3 | 9 | 12

3. Other Pre Specified Outcome: Median Cumulative Number of CD34+ Cells Collected During Apheresis
Description: Median cumulative total number of CD34+ cells collected during apheresis.
Time Frame: Days 5-8
Population: Participants who received at least one dose of plerixafor
Measure: Median (Full Range); unit: CD34+ cells (*10^6 / kg)
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 23 | 26 | 49
CD34+ cells (*10^6 / kg) | 5.2 [1.5 to 18.9] | 11.1 [4.4 to 22.5] | 5.9 [1.5 to 22.5]

4. Secondary Outcome: Number of Transplants in Which Participants Achieved Polymorphonuclear Leukocyte (PMN) Engraftment by Day 12 But No Later Than Day 21 Post Peripheral Blood Stem Cell (PBSC) Transplant
Description: Participants were monitored for polymorphonuclear leukocyte (PMN) engraftment as per the local standard of care. The target for engraftment was 12 days after PBSC transplant and no transplant taking longer than 21 days for engraftment.
Time Frame: 2 months
Population: Participants who received a transplant. Two participants in the MM group received a second transplant.
Measure: Number; unit: number of transplants
Units Other Than Participants: transplants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 22 | 25 | 47
Number analyzed (transplants) | 22 | 27 | 49
number of transplants
  ≤ Day 12 | 19 | 20 | 39
  Day 13 to Day 21 | 3 | 7 | 10
  ≥ Day 22 | 0 | 0 | 0

5. Other Pre Specified Outcome: Number of Transplants in Which Participants Achieved Platelet (PLT) Engraftment by Day 12 But No Later Than Day 21 Post Peripheral Blood Stem Cell (PBSC) Transplant
Description: Participants were monitored for platelet (PLT) engraftment as per the local standard of care. The target for engraftment was 12 days after PBSC transplant and no transplant taking longer than 21 days for engraftment.
Time Frame: 2 months
Population: A total of 47 participants were transplanted. Two participants in the MM group received a second transplant using cells collected on study. One participant in the MM group did not have PLT engraftment information recorded, however did report a durable graft at month 12 post transplant.
Measure: Number; unit: number of transplants
Units Other Than Participants: transplants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 22 | 24 | 46
Number analyzed (transplants) | 22 | 26 | 48
number of transplants
  ≤ Day 12 | 7 | 7 | 14
  Day 13 to Day 21 | 10 | 18 | 28
  ≥ Day 22 | 5 | 1 | 6

6. Other Pre Specified Outcome: Number of Participants With Durable Engraftment 12 Months After Transplantation
Description: The number of participants maintaining a durable graft 12 months after autologous transplantation. A durable graft is defined as the maintenance of normal blood counts.
Time Frame: Approximately 13 months (12 months post-transplant )
Population: Participants who received plerixafor, underwent transplantation, and were evaluable 12 months post transplant. The one participant who did not have a durable graft at 12 months had received chemotherapy for relapse approximately 9 months after transplantation.
Measure: Number; unit: participants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 21 | 23 | 44
participants | 21 | 22 | 43

ADVERSE EVENTS:
Time Frame: First day of G-CSF administration to the day prior to chemotherapy/ablative treatment in preparation of first transplant. This period includes the G-CSF, plerixafor treatment and rest period.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Each AE table includes events, regardless of reported relationship to study treatment or grade.
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/26
Other Adverse Events (participants affected / at risk) | 23/23 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL) (N=23) | Multiple Myeloma (MM) (N=26)
Heparin-induced thrombocytopenia (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL) (N=23) | Multiple Myeloma (MM) (N=26)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3
Palpitations (Cardiac disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 13 | 10
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 8
Oral pain (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 3
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Catheter related complication (General disorders) | 1 | 1
Catheter site discharge (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 2 | 1
Catheter site pain (General disorders) | 2 | 0
Catheter site pruritus (General disorders) | 0 | 1
Catheter site related reaction (General disorders) | 0 | 2
Catheter thrombosis (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 7 | 4
Feeling cold (General disorders) | 0 | 1
Hunger (General disorders) | 2 | 0
Injection site erythema (General disorders) | 6 | 3
Injection site haemorrhage (General disorders) | 2 | 0
Injection site irritation (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 1
Injection site swelling (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 1
Secretion discharge (General disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Blood stem cell harvest failure (Injury, poisoning and procedural complications) | 1 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Bacteria stool identified (Investigations) | 0 | 1
Blood alkaline phosphatase decreased (Investigations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0
Heart rate irregular (Investigations) | 1 | 0
Lymphocyte count abnormal (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 9 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 6
Nervousness (Psychiatric disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.